CLINICAL TRIAL: NCT02674568
Title: An Open-label, Single-Arm, Phase 2 Study Evaluating the Efficacy, Safety and Pharmacokinetics of Rovalpituzumab Tesirine (SC16LD6.5) for Third-line and Later Treatment of Subjects With Relapsed or Refractory Delta-Like Protein 3-Expressing Small Cell Lung Cancer (TRINITY)
Brief Title: Study of Rovalpituzumab Tesirine (SC16LD6.5) for Third-Line and Later Treatment of Subjects With Relapsed or Refractory Delta-Like Protein 3-Expressing Small Cell Lung Cancer
Acronym: TRINITY
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCRX001-002; 2015-004506-42 (EudraCT Number)
Record Dates: First submitted 2016-01-29; First posted 2016-02-04 (Estimated); Results first posted 2019-10-23 (Actual); Last update posted 2021-07-30 (Actual); Status verified 2021-07

CONDITIONS: Small Cell Lung Cancer
Keywords: SCLC; Small Cell Lung Cancer; DLL#; Relapsed; Refractory
MeSH Terms: conditions — Small Cell Lung Carcinoma; Recurrence | interventions — rovalpituzumab tesirine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Rovalpituzumab Tesirine (Experimental): 0.3 mg/kg rovalpituzumab tesirine administered intravenously on Day 1 of each 42-day cycle (every 6 weeks; Q6W) for 2 cycles. An additional 2 cycles of rovalpituzumab tesirine (retreatment) was permitted for eligible participants.
  Interventions: Drug: Rovalpituzumab tesirine

INTERVENTIONS:
Drug: Rovalpituzumab tesirine — Rovalpituzumab tesirine is a DLL3 targeted antibody drug conjugate (ADC).
  Other Names: SC16LD6.5

SUMMARY:
The purpose of this study is to determine the efficacy of rovalpituzumab tesirine as a third-line and later treatment for participants with relapsed or refractory delta-like protein 3 (DLL3) expressing small cell lung cancer (SCLC).

ELIGIBILITY:
Inclusion Criteria:

1. Adult aged 18 years or older
2. Histologically confirmed SCLC with documented disease progression after at least 2 prior systemic regimens, including at least one platinum-based regimen
3. DLL3-expressing SCLC based on central immunohistochemistry (IHC) assessment of banked or otherwise representative tumor tissue. Positive is defined as staining in ≥ 1% of tumor cells
4. Measurable disease as defined by Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1
5. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
6. Minimum life expectancy of at least 12 weeks
7. Subjects with a history of central nervous system (CNS) metastases must have documentation of stable or improved status based on brain imaging for at least 2 weeks after completion of definitive treatment and within 2 weeks prior to first dose of study drug, off or on a stable dose of corticosteroids
8. Recovery to Grade 1 of any clinically significant toxicity (excluding alopecia) prior to initiation of study drug administration
9. Adequate hematologic and organ function as confirmed by laboratory values
10. Last dose of any prior therapy administered by the following time intervals before the first dose of study drug:

    * Chemotherapy, small molecule inhibitors, radiation, and/or other investigational anticancer agents (excluding investigational monoclonal antibodies): 2 weeks
    * Immune-checkpoint inhibitors (i.e., anti-PD-1, anti-PD-L1, or anti-CTLA-4): 4 weeks
    * Other monoclonal antibodies, antibody-drug conjugates, radioimmunoconjugates, or T-cell or other cell-based therapies: 4 weeks (2 weeks with documented disease progression)
11. Females of childbearing potential must have a negative beta human chorionic gonadotropin (β-hCG) pregnancy test result within 7 days prior to the first dose of study drug. Females of non-childbearing potential are those who are postmenopausal greater than 1 year or who have had a bilateral tubal ligation or hysterectomy.

Exclusion Criteria:

1. Any significant medical condition, including any suggested by screening laboratory findings that, in the opinion of the investigator or sponsor, may place the subject at undue risk from the study, including but not necessarily limited to uncontrolled hypertension and/or diabetes, clinically significant pulmonary disease (e.g., chronic obstructive pulmonary disease requiring hospitalization within 6 months) or neurological disorder (e.g., seizure disorder active within 6 months)
2. Documented history of a cerebral vascular event (stroke or transient ischemic attack), unstable angina, myocardial infarction, or cardiac symptoms consistent with New York Heart Association (NYHA) Class III-IV within 6 months prior to their first dose of study drug
3. Recent or ongoing serious infection, including:

   * Any active grade 3 or higher (per National Cancer Institute's Common Terminology Criteria for Adverse Events [NCI CTCAE] version 4.03) viral, bacterial, or fungal infection within 2 weeks of the first dose of the study drug. Routine antimicrobial prophylaxis is permitted.
   * Known seropositivity for or active infection by human immunodeficiency virus (HIV)
   * Active Hepatitis B (by surface antigen expression or polymerase chain reaction) or C (by polymerase chain reaction) infection or on hepatitis-related antiviral therapy within 6 months of first dose of study drug.
4. Women who are breastfeeding
5. Systemic therapy with corticosteroids at >20 mg/day prednisone or equivalent within 1 week prior to the first dose of study drug
6. History of another invasive malignancy that has not been in remission for at least 3 years. Exceptions to the 3 year limit include nonmelanoma skin cancer, curatively treated localized prostate cancer, and cervical cancer in situ on biopsy or squamous intraepithelial lesion on pap smear
7. Prior exposure to a pyrrolobenzodiazepine (PBD)-based drug, or known hypersensitivity to rovalpituzumab tesirine or excipient contained in the drug formulation, unless undergoing retreatment with rovalpituzumab tesirine in the context of this protocol

Min Age: 18 Years | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 342 (Actual)
Dates: Start 2016-01-25 (Actual); Primary Completion 2018-10-19 (Actual); Study Completion 2018-10-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: AbbVie Inc., Study Director — AbbVie

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible data sharing regarding the clinical trials we sponsor. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information (e.g., protocols and clinical study reports), as long as the trials are not part of an ongoing or planned regulatory submission. This includes requests for clinical trial data for unlicensed products and indications.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data requests can be submitted at any time and the data will be accessible for 12 months, with possible extensions considered.
Access Criteria: Access to this clinical trial data can be requested by any qualified researchers who engage in rigorous, independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Sharing Agreement (DSA). For more information on the process, or to submit a request, visit the following link.
URL: https://www.abbvie.com/our-science/clinical-trials/clinical-trials-data-and-information-sharing/data-and-information-sharing-with-qualified-researchers.html

REFERENCES:
- [Background] Morgensztern D, Besse B, Greillier L, Santana-Davila R, Ready N, Hann CL, Glisson BS, Farago AF, Dowlati A, Rudin CM, Le Moulec S, Lally S, Yalamanchili S, Wolf J, Govindan R, Carbone DP. Efficacy and Safety of Rovalpituzumab Tesirine in Third-Line and Beyond Patients with DLL3-Expressing, Relapsed/Refractory Small-Cell Lung Cancer: Results From the Phase II TRINITY Study. Clin Cancer Res. 2019 Dec 1;25(23):6958-6966. doi: 10.1158/1078-0432.CCR-19-1133. Epub 2019 Sep 10. PMID 31506387

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 342 participants were enrolled; 3 participants were not dosed.
Period: Overall Study
Arm/Group | Rovalpituzumab Tesirine
Started | 339 (Enrolled and dosed.)
Delta-like Protein 3 (DLL3) High (DLL3 High Participants: tumors with ≥75% of cells expressing DLL3 are classified as "DLL3 high") | 238
DLL3 Positive (DLL3 Positive Participants: tumors with ≥25% cells expressing DLL3 are classified as "DLL3 positive") | 287
Completed ('Completed'=still on study; 'Not Completed'=discontinued study) | 0
Not Completed | 339
Not completed — Withdrawal by Subject | 5
Not completed — Death | 303
Not completed — Physician Decision | 2
Not completed — Lost to Follow-up | 9
Not completed — Other, Not Specified | 20

BASELINE CHARACTERISTICS:
Groups:
- Rovalpituzumab Tesirine: 0.3 mg/kg rovalpituzumab tesirine administered intravenously on Day 1 of each 42-day cycle (Q6W) for 2 cycles. An additional 2 cycles of rovalpituzumab tesirine (retreatment) was permitted for eligible participants.
Arm/Group | Rovalpituzumab Tesirine
Number analyzed (Participants) | 339
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.9 (9.36)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 169
  Male | 170
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10
  Not Hispanic or Latino | 272
  Unknown or Not Reported | 57
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 11
  White | 265
  More than one race | 3
  Unknown or Not Reported | 56

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate
Description: Objective response is defined as a participant with the best overall response of complete response (CR) or partial response (PR), per Response Evaluation Criteria in Solid Tumors (RECIST) v 1.1, prior to receiving any subsequent anticancer therapy and retreatment, and is confirmed by a consecutive response assessment at least 4 weeks (28 days) from the initial determination of CR/PR. Analyzed based on response assessments from both the Independent Review Committee (IRC) and investigators.
  CR: disappearance of all target lesions.Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm.
  PR: at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: up to 122.4 weeks; mean (SD) duration of follow-up was 29.0 (23.77) weeks
Population: Modified Intent to Treat Population: all participants who received any amount of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Rovalpituzumab Tesirine: DLL3 High: 'DLL3 High' (tumors with ≥75% of cells expressing DLL3) participants received 0.3 mg/kg rovalpituzumab tesirine administered intravenously on Day 1 of each 42-day cycle (Q6W) for 2 cycles. An additional 2 cycles of rovalpituzumab tesirine (retreatment) was permitted for eligible participants.
- Rovalpituzumab Tesirine: DLL3 Positive: 'DLL3 Positive' (tumors with ≥25% of cells expressing DLL3) participants received 0.3 mg/kg rovalpituzumab tesirine administered intravenously on Day 1 of each 42-day cycle (Q6W) for 2 cycles. An additional 2 cycles of rovalpituzumab tesirine (retreatment) was permitted for eligible participants.
Arm/Group | Rovalpituzumab Tesirine: DLL3 High | Rovalpituzumab Tesirine: DLL3 Positive
Number analyzed (Participants) | 238 | 287
percentage of participants
  IRC | 15.5 [11.2 to 20.8] | 14.6 [10.8 to 19.3]
  Investigator | 19.3 [14.5 to 24.9] | 18.8 [14.5 to 23.8]

2. Primary Outcome: Overall Survival
Description: Overall survival is defined as the time from the first dose date to death for any reason. Participants who were alive at the clinical data cut-off were censored at the last known alive date. Based on Kaplan-Meier estimates.
Time Frame: up to 122.4 weeks; mean (SD) duration of follow-up was 29.0 (23.77) weeks
Population: Modified Intent to Treat Population: all participants who received any amount of study drug.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Rovalpituzumab Tesirine: DLL3 High | Rovalpituzumab Tesirine: DLL3 Positive
Number analyzed (Participants) | 238 | 287
months | 5.3 [4.7 to 5.8] | 5.3 [4.7 to 5.8]

3. Secondary Outcome: Overall Response Rate
Description: Overall response rate is defined as the percentage of participants with a response of CR or PR, regardless of confirmation, per RECIST v 1.1 prior to receiving any subsequent anticancer therapy and retreatment. Any participants not exhibiting a response (CR or PR) as defined above were considered non-responders. Analyzed based on response assessments from both the IRC and investigators.
  CR: disappearance of all target lesions.Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm.
  PR: at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: up to 122.4 weeks; mean (SD) duration of follow-up was 29.0 (23.77) weeks
Population: Modified Intent to Treat Population: all participants who received any amount of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Rovalpituzumab Tesirine: DLL3 High | Rovalpituzumab Tesirine: DLL3 Positive
Number analyzed (Participants) | 238 | 287
percentage of participants
  IRC | 23.1 [17.9 to 29.0] | 22.0 [17.3 to 27.2]
  Investigator | 26.9 [21.4 to 33.0] | 25.8 [20.8 to 31.3]

4. Secondary Outcome: Duration of Objective Response
Description: Duration of objective response is defined as the time from the date of first documented CR or PR of participants with a confirmed response to the documented date of progressive disease (PD) or death, whichever occurred first. Participants who neither progressed nor died are censored at the last evaluable disease assessment. Analyzed based on response assessments from both the IRC and investigators. Based on Kaplan-Meier estimates.
  CR: disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm.
  PR: at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
  PD: at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (includes the baseline sum). The sum must also demonstrate an absolute increase of at least 5 mm. (The appearance of one or more new lesions is also considered progression.)
Time Frame: up to 122.4 weeks; mean (SD) duration of follow-up was 29.0 (23.77) weeks
Population: Modified Intent to Treat Population: all participants who received any amount of study drug and had an objective response.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Rovalpituzumab Tesirine: DLL3 High | Rovalpituzumab Tesirine: DLL3 Positive
Number analyzed (Participants) | 46 | 54
months
  IRC: number analyzed (Participants) | 37 | 42
  IRC | 4.0 [3.0 to 4.2] | 4.1 [3.0 to 4.2]
  Investigator | 4.0 [2.9 to 4.2] | 4.0 [2.9 to 4.3]

5. Secondary Outcome: Progression-Free Survival
Description: Progression-free survival is defined as the time from the first dose date to the documented date of PD or death, whichever occurred first. Participants who neither progressed nor died were censored at the last evaluable disease assessment. Analyzed based on response assessments from both the IRC and investigators. Based on Kaplan-Meier estimates.
  PD: at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (includes the baseline sum). The sum must also demonstrate an absolute increase of at least 5 mm. (The appearance of one or more new lesions is also considered progression.)
Time Frame: up to 122.4 weeks; mean (SD) duration of follow-up was 29.0 (23.77) weeks
Population: Modified Intent to Treat Population: all participants who received any amount of study drug.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Rovalpituzumab Tesirine: DLL3 High | Rovalpituzumab Tesirine: DLL3 Positive
Number analyzed (Participants) | 238 | 287
months
  IRC | 3.8 [3.3 to 4.1] | 3.8 [3.3 to 4.0]
  Investigator | 3.9 [3.3 to 4.1] | 3.9 [3.3 to 4.0]

6. Secondary Outcome: Clinical Benefit Rate
Description: Clinical benefit rate is defined as the percentage of participants with an overall response of CR or PR or stable disease (SD) with SD of a minimum duration of 42 days from the first dose date. Analyzed based on response assessments from both the IRC and investigators.
  CR: disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm.
  PR: at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
  SD: neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study.
  PD: at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (includes the baseline sum). The sum must also demonstrate an absolute increase of at least 5 mm. (The appearance of one or more new lesions is also considered progression.)
Time Frame: up to 122.4 weeks; mean (SD) duration of follow-up was 29.0 (23.77) weeks
Population: Modified Intent to Treat Population: all participants who received any amount of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Rovalpituzumab Tesirine: DLL3 High | Rovalpituzumab Tesirine: DLL3 Positive
Number analyzed (Participants) | 238 | 287
percentage of participants
  IRC | 73.9 [67.9 to 79.4] | 72.1 [66.6 to 77.2]
  Investigator | 71.0 [64.8 to 76.7] | 68.6 [62.9 to 74.0]

7. Secondary Outcome: Duration of Clinical Benefit
Description: Duration of clinical benefit is defined as time from the date of first documented CR or PR or SD of ≥ 42 days from first dose date (-7 days to allow for scheduled visit window per the protocol) to the documented date PD or death, whichever occurs first. Analyzed based on response assessments from both the IRC and investigators.
  CR: disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm.
  PR: at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
  SD: neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study.
Time Frame: up to 122.4 weeks; mean (SD) duration of follow-up was 29.0 (23.77) weeks
Population: Modified Intent to Treat Population: all participants who received any amount of study drug with best overall response of CR or PR or SD.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Rovalpituzumab Tesirine: DLL3 High | Rovalpituzumab Tesirine: DLL3 Positive
Number analyzed (Participants) | 176 | 207
months
  IRC | 2.9 [2.8 to 3.2] | 2.9 [2.8 to 3.0]
  Investigator: number analyzed (Participants) | 169 | 197
  Investigator | 3.0 [2.9 to 3.3] | 3.0 [2.9 to 3.2]

8. Secondary Outcome: Rovalpituzumab Tesirine Antibody-Drug Conjugate Plasma Concentrations by Study Visit
Time Frame: Cycle 1: Day 1, 30 minutes pre-infusion; Day 1, 30 minutes post-infusion; Day 3; Day 15; Day 29. Cycle 2: Day 1, 30 minutes pre-infusion; Day 1, 30 minutes post-infusion; Day 3; Day 15; Day 29; End of Treatment (up to Day 29).
Population: Pharmacokinetic Analysis Population: all participants who receive at least 1 dose of study treatment and at least 1 post-baseline blood sample following a dose of study treatment and had an assessment at given time point.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Rovalpituzumab Tesirine: Initial Treatment Period: 0.3 mg/kg rovalpituzumab tesirine administered intravenously on Day 1 of each 42-day cycle (Q6W) for 2 cycles.
- Rovalpituzumab Tesirine: Re-Treatment 1: 0.3 mg/kg rovalpituzumab tesirine administered intravenously on Day 1 of retreatment Cycle 1
- Rovalpituzumab Tesirine: Re-Treatment 2: 0.3 mg/kg rovalpituzumab tesirine administered intravenously on Day 1 of retreatment Cycle 2
Arm/Group | Rovalpituzumab Tesirine: Initial Treatment Period | Rovalpituzumab Tesirine: Re-Treatment 1 | Rovalpituzumab Tesirine: Re-Treatment 2
Number analyzed (Participants) | 329 | 20 | 2
ng/mL
  Cycle 1: Day 1, 30 minutes pre-infusion | 180.9 (1215.03) | 236.6 (923.44) | 148.2 (81.81)
  Cycle 1: Day 1, 30 minutes post-infusion | 7611.6 (1980.49) | 6365.5 (1763.08) | 6690.0 (2050.61)
  Cycle 1: Day 3: number analyzed (Participants) | 317 | 20 | 2
  Cycle 1: Day 3 | 4535.2 (1398.49) | 3740.5 (1454.87) | 4630.0 (1866.76)
  Cycle 1: Day 15: number analyzed (Participants) | 300 | 15 | 2
  Cycle 1: Day 15 | 1472.8 (573.90) | 1323.3 (504.33) | 1390.0 (381.84)
  Cycle 1: Day 29: number analyzed (Participants) | 279 | 18 | 2
  Cycle 1: Day 29 | 816.3 (379.15) | 793.8 (322.90) | 956.5 (61.52)
  Cycle 2: Day 1, 30 minutes pre-infusion: number analyzed (Participants) | 223 | 15 | 1
  Cycle 2: Day 1, 30 minutes pre-infusion | 532.2 (592.90) | 518.6 (226.45) | 601.0 (NA) — 1 participant was analyzed.
  Cycle 2: Day 1, 30 minutes post-infusion: number analyzed (Participants) | 216 | 15 | 1
  Cycle 2: Day 1, 30 minutes post-infusion | 7535.6 (1928.74) | 6602.7 (1508.23) | 7880.0 (NA) — 1 participant was analyzed.
  Cycle 2: Day 3: number analyzed (Participants) | 205 | 13 | 1
  Cycle 2: Day 3 | 4791.1 (1373.70) | 4670.8 (1539.65) | 3840.0 (NA) — 1 participant was analyzed.
  Cycle 2: Day 15: number analyzed (Participants) | 206 | 13 | 1
  Cycle 2: Day 15 | 1845.5 (688.47) | 1857.7 (599.65) | 2030.0 (NA) — 1 participant was analyzed.
  Cycle 2: Day 29: number analyzed (Participants) | 175 | 14 | 1
  Cycle 2: Day 29 | 1029.3 (362.28) | 1077.7 (362.33) | 1300.0 (NA) — 1 participant was analyzed.
  End of Treatment: number analyzed (Participants) | 213 | 15 | 2
  End of Treatment | 558.5 (296.09) | 686.9 (354.68) | 679.5 (64.35)

9. Secondary Outcome: Number of Anti-Therapeutic Antibody (ATA) Positive Participants
Time Frame: up to 122.4 weeks; mean (SD) duration of follow-up was 29.0 (23.77) weeks
Population: All participants who received rovalpituzumab tesirine and had at least one sample screened for ATA against rovalpituzumab tesirine antibody-drug conjugate concentration.
Measure: Count of Participants; unit: Participants
Arm/Group | Rovalpituzumab Tesirine
Number analyzed (Participants) | 336
Participants
  Positive at Any Study Visit | 11
  Positive After First Dose of Study Drug: number analyzed (Participants) | 276
  Positive After First Dose of Study Drug | 3

10. Secondary Outcome: Number of Participants With Treatment-Related Adverse Events (TEAEs) During Initial Treatment
Description: An adverse event (AE) is defined as any untoward medical occurrence which does not necessarily have a causal relationship with this treatment. A serious adverse event (SAE) is any untoward medical occurrence that at any dose: is fatal or life-threatening; results in death or hospitalization; is disabling/incapacitating or a congenital anomaly/birth defect; is medically significant. AE severity was graded using the National Cancer Institute's Common Terminology Criteria for Adverse Events (NCI CTCAE), version 4.03 terminology: grade 1=mild; grade 2=moderate; grade 3=severe; grade 4 life-threatening; grade 5=death. TEAEs were defined as AEs that were newly occurring or worsened following study treatment.
Time Frame: From first dose of study drug through the end of the initial treatment period (84 ± 6 days)
Population: Safety analysis population: all participants who received any amount of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Rovalpituzumab Tesirine
Number analyzed (Participants) | 339
Participants
  Any TEAE | 335
  Treatment Emergent SAE | 171
  TEAE Maximum Severity Grade 3/4 | 179
  TEAE Leading to Drug WIthdrawal | 25
  TEAE Leading to Dose Interruption | 33
  TEAE Leading to Dose Reduction | 32
  TEAE Reasonably Possibly Related to Study Drug | 308
  Fatal AE | 34

11. Secondary Outcome: Number of Participants With TEAEs Occurring in at Least 10% of All Participants During Initial Treatment
Description: TEAEs were defined as AEs that were newly occurring or worsened following study treatment.
Time Frame: From first dose of study drug through the end of the initial treatment period (84 ± 6 days)
Population: Safety analysis population: all participants who received any amount of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Rovalpituzumab Tesirine
Number analyzed (Participants) | 339
Participants
  Any TEAE | 335
  Fatigue | 129
  Photosensitivity Reaction | 123
  Pleural effusion | 113
  Oedema peripheral | 105
  Decreased appetite | 102
  Nausea | 88
  Dyspnoea | 83
  Thrombocytopenia | 83
  Constipation | 75
  Vomiting | 59
  Anaemia | 58
  Cough | 54
  Hypoalbuminaemia | 52
  Pericardial effusion | 50
  Abdominal pain | 50
  Asthenia | 50
  Diarrhoea | 47

ADVERSE EVENTS:
Time Frame: From first dose of study drug through the end of treatment (EOT; 42 ± 3 days after last dose, or within 7 days of documentation of the decision to discontinue treatment, whichever was later) or 30 days after last study treatment, whichever was later. Mean (SD) duration of follow-up (ie, from the first dose date to the last known date alive or death date) was 29.0 (23.77) weeks.
Arm/Group | Rovalpituzumab Tesirine
All-Cause Mortality (participants affected / at risk) | 303/339
Serious Adverse Events (participants affected / at risk) | 178/339
Other Adverse Events (participants affected / at risk) | 322/339
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rovalpituzumab Tesirine (N=339)
Anaemia (Blood and lymphatic system disorders) | 7 (7)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 11 (13)
Atrial fibrillation (Cardiac disorders) | 6 (6)
Cardiac arrest (Cardiac disorders) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 1 (1)
Cardiac tamponade (Cardiac disorders) | 4 (4)
Cardiopulmonary failure (Cardiac disorders) | 1 (2)
Pericardial effusion (Cardiac disorders) | 14 (19)
Sinus bradycardia (Cardiac disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 9 (10)
Ascites (Gastrointestinal disorders) | 4 (4)
Colitis (Gastrointestinal disorders) | 2 (2)
Constipation (Gastrointestinal disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 1 (2)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1)
Intestinal ischaemia (Gastrointestinal disorders) | 1 (2)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 7 (8)
Pancreatitis (Gastrointestinal disorders) | 2 (2)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Asthenia (General disorders) | 4 (6)
Fatigue (General disorders) | 5 (5)
Gait disturbance (General disorders) | 1 (1)
General physical health deterioration (General disorders) | 8 (14)
Generalised oedema (General disorders) | 8 (10)
Oedema peripheral (General disorders) | 8 (10)
Pain (General disorders) | 3 (4)
Pyrexia (General disorders) | 3 (3)
Cholangitis (Hepatobiliary disorders) | 1 (1)
Drug-induced liver injury (Hepatobiliary disorders) | 1 (2)
Hepatic pain (Hepatobiliary disorders) | 1 (1)
Hepatocellular injury (Hepatobiliary disorders) | 3 (4)
Hepatotoxicity (Hepatobiliary disorders) | 2 (2)
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 (2)
Bacterial infection (Infections and infestations) | 1 (1)
Bronchitis (Infections and infestations) | 2 (2)
Cellulitis (Infections and infestations) | 1 (1)
Cerebral toxoplasmosis (Infections and infestations) | 1 (1)
Clostridium difficile colitis (Infections and infestations) | 2 (3)
Device related infection (Infections and infestations) | 1 (1)
Diverticulitis (Infections and infestations) | 1 (1)
Infection (Infections and infestations) | 1 (1)
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 1 (1)
Lung infection (Infections and infestations) | 1 (1)
Oesophageal candidiasis (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 12 (16)
Pulmonary sepsis (Infections and infestations) | 1 (1)
Respiratory tract infection (Infections and infestations) | 3 (4)
Sepsis (Infections and infestations) | 6 (8)
Septic shock (Infections and infestations) | 1 (2)
Urinary tract infection (Infections and infestations) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 1 (1)
Humerus fracture (Injury, poisoning and procedural complications) | 1 (1)
Ligament sprain (Injury, poisoning and procedural complications) | 1 (1)
Pneumonitis chemical (Injury, poisoning and procedural complications) | 1 (2)
Tracheal haemorrhage (Injury, poisoning and procedural complications) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (2)
Blood uric acid increased (Investigations) | 1 (1)
Ejection fraction decreased (Investigations) | 1 (1)
Liver function test increased (Investigations) | 2 (2)
Platelet count decreased (Investigations) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 2 (2)
Hyponatraemia (Metabolism and nutrition disorders) | 6 (6)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Flank pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Spinal pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (2)
Metastases to pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Metastasis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Hemiparesis (Nervous system disorders) | 1 (1)
Seizure (Nervous system disorders) | 1 (1)
Spinal cord compression (Nervous system disorders) | 2 (2)
Device occlusion (Product Issues) | 1 (1)
Confusional state (Psychiatric disorders) | 5 (5)
Delirium (Psychiatric disorders) | 2 (2)
Disorientation (Psychiatric disorders) | 1 (1)
Mental status changes (Psychiatric disorders) | 4 (4)
Acute kidney injury (Renal and urinary disorders) | 3 (3)
Haematuria (Renal and urinary disorders) | 1 (1)
Renal failure (Renal and urinary disorders) | 1 (1)
Renal impairment (Renal and urinary disorders) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 49 (62)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 (5)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 7 (11)
Tracheal stenosis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dermatitis exfoliative (Skin and subcutaneous tissue disorders) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1)
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 6 (7)
Capillary leak syndrome (Vascular disorders) | 2 (2)
Deep vein thrombosis (Vascular disorders) | 2 (2)
Haemorrhage (Vascular disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
Intermittent claudication (Vascular disorders) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 1 (1)
Peripheral ischaemia (Vascular disorders) | 1 (1)
Superior vena cava syndrome (Vascular disorders) | 3 (3)
Venous thrombosis limb (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Rovalpituzumab Tesirine (N=339)
Anaemia (Blood and lymphatic system disorders) | 54 (88)
Thrombocytopenia (Blood and lymphatic system disorders) | 73 (140)
Pericardial effusion (Cardiac disorders) | 38 (40)
Abdominal distension (Gastrointestinal disorders) | 20 (21)
Abdominal pain (Gastrointestinal disorders) | 42 (59)
Constipation (Gastrointestinal disorders) | 74 (87)
Diarrhoea (Gastrointestinal disorders) | 46 (50)
Nausea (Gastrointestinal disorders) | 82 (101)
Vomiting (Gastrointestinal disorders) | 60 (75)
Asthenia (General disorders) | 48 (81)
Face oedema (General disorders) | 32 (32)
Fatigue (General disorders) | 125 (170)
Non-cardiac chest pain (General disorders) | 19 (21)
Oedema peripheral (General disorders) | 101 (136)
Urinary tract infection (Infections and infestations) | 27 (32)
Alanine aminotransferase increased (Investigations) | 20 (33)
Aspartate aminotransferase increased (Investigations) | 20 (27)
Weight decreased (Investigations) | 32 (36)
Decreased appetite (Metabolism and nutrition disorders) | 104 (124)
Dehydration (Metabolism and nutrition disorders) | 19 (22)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 54 (70)
Hypokalaemia (Metabolism and nutrition disorders) | 19 (23)
Back pain (Musculoskeletal and connective tissue disorders) | 30 (36)
Myalgia (Musculoskeletal and connective tissue disorders) | 22 (27)
Dizziness (Nervous system disorders) | 33 (37)
Headache (Nervous system disorders) | 18 (18)
Insomnia (Psychiatric disorders) | 26 (26)
Cough (Respiratory, thoracic and mediastinal disorders) | 56 (67)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 83 (107)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 69 (84)
Dry skin (Skin and subcutaneous tissue disorders) | 25 (28)
Erythema (Skin and subcutaneous tissue disorders) | 30 (37)
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 119 (199)
Rash (Skin and subcutaneous tissue disorders) | 26 (30)
Hypotension (Vascular disorders) | 19 (21)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.

DOCUMENTS (2):
  • Study Protocol (2016-11-18): https://cdn.clinicaltrials.gov/large-docs/68/NCT02674568/Prot_000.pdf
  • Statistical Analysis Plan (2018-02-14): https://cdn.clinicaltrials.gov/large-docs/68/NCT02674568/SAP_001.pdf